CLINICAL TRIAL: NCT00509964
Title: A Randomized Phase II Trial of Irinotecan Monotherapy Versus Irinotecan, Leucovorin and 5-FU (ILF) Combination Chemotherapy in Patients With Advanced Gastric Cancer Failing Prior Chemotherapy
Brief Title: Second-Line Irinotecan vs. ILF for AGC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMO-GI-71
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Stomach Neoplasm; Metastatic; Second-Line
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will receive irinotecan 150 mg/m2 intravenously on day 1 every 2 weeks.
  Interventions: Drug: irinotecan
- 2 (Active Comparator): Patients will receive irinotecan 150 mg/m2 intravenously, in combination with leucovorin and infusional 5-fluorouracil, on day 1 every 2 weeks.
  Interventions: Drug: ILF

INTERVENTIONS:
Drug: irinotecan — Patients will receive irinotecan 150 mg/m2 intravenously on day 1 every 2 weeks.
  Arms: 1
Drug: ILF — Patients will receive irinotecan 150 mg/m2 intravenously, in combination with leucovorin and 5-fluorouracil, on day 1 every 2 weeks.
  Arms: 2

SUMMARY:
Patients with recurrent or metastatic gastric cancer can benefit from palliative chemotherapy. However, over half of patients with metastatic gastric cancer who received chemotherapy failed to achieve response and even in these responders, the duration of responses was as short as a few months. Patients with metastatic gastric cancer who fail to respond or have relapse after first line chemotherapy have a grim prognosis and a standard salvage treatment is not available.

We designed this phase II trial to determine the efficacy and safety of irinotecan monotherapy or combination (ILF) as second-line therapy for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed gastric cancer
* inoperable, recurrent, or metastatic
* performance status 0 to 2
* failed after one or more prior chemotherapy for advanced disease
* informed consent

Exclusion Criteria:

* active infection
* severe co-morbidities
* previously treated with irinotecan or similar drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-05; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, Incheon, South Korea